CLINICAL TRIAL: NCT00732992
Title: Phase 1 Study Of Sunitinib (SU011248) In Combination With Pemetrexed In Patients With Advanced Solid Malignancies In Japan
Brief Title: A Safety Study Of Sunitinib In Combination With Pemetrexed In Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181165
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Neoplasm, Malignant
Keywords: Solid tumor; malignancy; sunitinib; pemetrexed; phase 1; neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Sunitinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDD (Experimental)
  Interventions: Drug: Sunitinib, Pemetrexed
- 2/1 (Experimental)
  Interventions: Drug: Sunitinib, Pemetrexed

INTERVENTIONS:
Drug: Sunitinib, Pemetrexed — Sunitinib daily by oral capsule in a continuous daily dosing regimen with pemetrexed every 3 weeks until progression or unacceptable toxicity.
  Other Names: Sutent, SU011248, Alimta
  Arms: CDD
Drug: Sunitinib, Pemetrexed — Sunitinib daily by oral capsule administered for 2 weeks out of every 3 weeks with pemetrexed every 3 weeks until progression or unacceptable toxicity.
  Other Names: Sutent, SU011248, Alimta
  Arms: 2/1

SUMMARY:
This study will assess if the combination of sunitinib and pemetrexed is tolerable when coadministered at each recommended dose/schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a solid malignancy that is refractory to standard therapy or for which no standard therapy exists.
* Patients has a good performance status (ECOG 0 or 1)

Exclusion Criteria:

* Prior treatment with either pemetrexed or SU011248.
* Coughing up blood within 4 weeks before starting study treatment (small amounts okey).
* Hypertension that cannot be controlled by medications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Osakasayama-shi, Osaka, Japan

REFERENCES:
- [Derived] Okamoto I, Shimizu T, Miyazaki M, Tsurutani J, Ichikawa Y, Terashima M, Takeda M, Fumita S, Ohki E, Kimura N, Hashimoto J, Nakagawa K. Feasibility study of two schedules of sunitinib in combination with pemetrexed in patients with advanced solid tumors. Invest New Drugs. 2012 Apr;30(2):639-46. doi: 10.1007/s10637-010-9565-5. Epub 2010 Oct 20. PMID 20960028

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib 37.5 mg/Day Continuous Daily Dosing: Sunitinib 37.5 mg was administered continuously on a daily basis. Pemetrexed 500 mg/m^2 was administered as intravenous infusion over 10 minutes on the first day (Day 1) of each 21-day cycle.
- Sunitinib 50 mg/Day Schedule-2/1: Sunitinib 50.0 mg was administered continuously on a daily basis for 2 weeks, followed by 1 week off treatment.
  Pemetrexed 500 mg/m^2 was administered as intravenous infusion over 10 minutes on the first day (Day 1) of each 21-day cycle.
Period: Overall Study
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing | Sunitinib 50 mg/Day Schedule-2/1
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Objective Progression or Relapse | 3 | 5
Not completed — Global Deterioration of Health Status | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing | Sunitinib 50 mg/Day Schedule-2/1 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Number; unit: Participants]
  20-44 years | 0 | 0 | 0
  45- 64 years | 4 | 2 | 6
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 4 | 10
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Score 0: Fully active, able to carry on all pre-disease performance without restriction; Score 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, such as light house work and office work.
  Participants
    Score 0 | 2 | 4 | 6
    Score 1 | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, adverse events graded as Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE) Grade 3 or higher , dose limiting toxicities (DLT), serious adverse events, adverse events resulted in discontinuation.
Time Frame: End of study (up to individual discontinuation)
Population: All subjects who received at least 1 dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing | Sunitinib 50 mg/Day Schedule-2/1
Number analyzed (Participants) | 6 | 6
Participants
  Any adverse events | 6 | 6
  Any dose limiting toxicities | 0 | 0
  Any serious adverse events | 2 | 1
  Any Grade-3 or -4 adverse events | 6 | 3
  Any Grade-5 adverse events (= death) | 0 | 0
  Discontinuation due to adverse events | 1 | 1

2. Secondary Outcome: Sunitinib Relative Dose Intensity in the "Sunitinib 37.5 mg/Day Continuous Daily Dosing" Treatment Arm
Description: Relative dose intensity was defined as percentage of total dose administered over total planned dose in the given period.
Time Frame: Up to Cycle 5 (end of study)
Population: Full analysis set = defined as "all enrolled patients". n = number of participants assessed for the relative dose intensity in the given period.
Measure: Median (Full Range); unit: percent of total planned dose
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 6
percent of total planned dose
  Cycle 1 (n=6) | 92.0 [75.9 to 100]
  Cycle 2 (n=6) | 54.8 [4.8 to 100]
  Cycle 3 (n=4) | 46.0 [14.9 to 95.2]
  Cycle 4 (n=4) | 55.6 [41.4 to 104.8]
  Cycle 5 (n=1) | 44.4 [44.4 to 44.4]

3. Secondary Outcome: Sunitinib Relative Dose Intensity in the "Sunitinib 50 mg/Day Schedule-2/1" Treatment Arm
Description: as for outcome 2
Time Frame: Up to Cycle 6
Population: as for outcome 2
Measure: Median (Full Range); unit: percent of total planned dose
Arm/Group | Sunitinib 50 mg/Day Schedule-2/1
Number analyzed (Participants) | 6
percent of total planned dose
  Cycle 1 (n=6) | 87.5 [60 to 100]
  Cycle 2 (n=5) | 80.4 [38.4 to 100]
  Cycle 3 (n=4) | 53.6 [42.9 to 75]
  Cycle 4 (n=3) | 50.0 [50 to 75]
  Cycle 5 (n=3) | 50.0 [41.1 to 50]
  Cycle 6 (n=3) | 50.0 [50 to 50]

4. Secondary Outcome: Trough and Maximum Concentration of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Description: Trough concentration was defined as observed concentration at 24 hours post dose. SU012662 is an active metabolite of sunitinib.
Time Frame: Cycle 2 Day 1: Pre-dose and 2, 4, 6, 8, 10, and 24 hours post-dose
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
nanogram/mL
  Sunitinib: Trough concentration | 45.6 (11.7)
  Sunitinib: Maximum concentration | 59.9 (10.9)
  SU012662: Trough concentration | 25.1 (5.08)
  SU012662: Maximum concentration | 31.6 (5.49)
  Total drug: Trough concentration | 70.6 (13.9)
  Total drug: Maximum concentration | 91.5 (14.2)

5. Secondary Outcome: AUC 0-24 of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Description: AUC0-24 = Area under the plasma concentration versus time curve to 24 hours post dose was calculated using the linear/logarithmic trapezoidal method. SU012662 is an active metabolite of sunitinib.
Time Frame: Cycle 2 Day 1: Pre-dose and 2, 4, 6, 8, 10, and 24 hours post-dose
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Mean (Standard Deviation); unit: nanogram*hour/mL
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
nanogram*hour/mL
  Sunitinib | 1190 (247)
  SU012662 | 675 (107)
  Total Drug | 1866 (269)

6. Secondary Outcome: Tmax of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Description: Tmax = Time to maximum plasma concentration. SU012662 is an active metabolite of sunitinib.
Time Frame: Cycle 2 Day 1: Pre-dose and 2, 4, 6, 8, 10, and 24 hours post-dose
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
hours
  Sunitinib | 4 [4 to 6]
  SU012662 | 4 [4 to 6]
  Total Drug | 4 [4 to 6]

7. Secondary Outcome: Maximum Concentration of Pemetrexed Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Time Frame: Cycle 2 Day 1: Pre-dose, 10 minutes after the start of infusion (immediately before the end of infusion), and 1, 2, 4, 6, 8, 10, and 24 hours post-dose
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
microgram/mL | 163 (30.7)

8. Secondary Outcome: AUC0-∞ of Pemetrexed Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Description: AUC0-∞ = Area under the plasma concentration versus time curve from zero time to infinity was calculated as the sum of AUClast and (Ct*/kel), where Ct* was the estimated concentration at the time of the last quantifiable concentration, kel was terminal phase rate constant that is estimated as the absolute value of the slope of a linear regression during the terminal phase of the natural-logarithm (ln) transformed concentration-time profile.
Time Frame: as for outcome 7
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Mean (Standard Deviation); unit: microgram*hour/mL
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
microgram*hour/mL | 191 (36.3)

9. Secondary Outcome: Terminal Phase Elimination Half-Life (T1/2) of Pemetrexed Following Continuous Daily Dosing of Sunitinib 37.5 mg/Day in Combination With Pemetrexed 500 mg/m^2 at Cycle 2 Day 1
Description: Terminal phase elimination half-life was calculated as "natural logarithm of 2 (ln2) divided by the rate constant for terminal phase (kel)".
Time Frame: as for outcome 7
Population: Participants who provided a plasma concentration data was included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing
Number analyzed (Participants) | 3
hours | 2.754 (0.531)

10. Secondary Outcome: Trough Concentrations of Sunitinib, SU012662, and Total Drug (Sunitinib + SU012662) After Coadministration of Sunitinib 50 mg/Day and Pemetrexed 500 mg/m^2 (Cycle 1 Day 1), Followed by Sunitinib 50 mg/Day on Schedule-2/1 at Cycle 1 Day 14 or 15
Description: as for outcome 4
Time Frame: Cycle 1 Day 14 (or 15): approximately 24 hours after the previous dose
Population: Participants who provided a plasma concentration data was included in the analysis
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | Sunitinib 50 mg/Day Schedule-2/1
Number analyzed (Participants) | 6
nanogram/mL
  Sunitinib | 78.5 (22.2)
  SU012662 | 38.2 (17.0)
  Total Drug | 117 (30.8)

11. Secondary Outcome: Summary of Best Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST): Number of Participants
Description: Complete response (CR): disappearance of all target lesions; Partial response (PR): >=30% decrease in the sum of the longest dimensions (SLD) of the target lesions taking as a reference the baseline SLD; Progressive disease (PD): >=20% increase in the SLD of the target lesions taking as a reference the smallest SLD recorded since the treatment started, or the appearance of >=1 new lesions; Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as a reference the smallest SLD since the treatment started.
Time Frame: End of study (Up to individual study discontinuation)
Population: Evaluable subjects = defined as all subjects who met all the following 3 requirements: 1) met the eligibility (inclusion and exclusion) criteria, 2) received at least 1 dose of the study drug, and 3) assessed appropriately at the baseline and had a measurable lesion based on the RECIST.
Measure: Number; unit: Participants
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing | Sunitinib 50 mg/Day Schedule-2/1
Number analyzed (Participants) | 4 | 4
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1 | 0
  Stable Disease (SD) | 2 | 3
  Progressive Disease (PD) | 1 | 1
  Not Evaluable (NE) | 0 | 0
  Objective Response (CR+PR) | 1 | 0
  Stable Disease (SD) >=184 days | 0 | 1
  Clinical Benefit (CR+PR+SD >=184 days) | 1 | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib 37.5 mg/Day Continuous Daily Dosing | Sunitinib 50 mg/Day Schedule-2/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg/Day Continuous Daily Dosing (N=6) | Sunitinib 50 mg/Day Schedule-2/1 (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg/Day Continuous Daily Dosing (N=6) | Sunitinib 50 mg/Day Schedule-2/1 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Chest pain (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 6
Influenza like illness (General disorders) | 0 | 1
Oedema (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 3
Folliculitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 3 | 2
Protein urine present (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 5 | 3
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.